CLINICAL TRIAL: NCT06709924
Title: Evaluating Effectiveness of Elevated Intra-abdominal Pressure (IAP) by PressureDOT
Acronym: IAP
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH113-REC2-139
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Intraabdominal Pressure
Keywords: Intraabdominal pressure; capsule
MeSH Terms: interventions — Exercise; Dosage Forms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Wrestling group: The ten participants who are expertise of wrestling and strong core muscle usage. After ingest the capsule, the signal transmission and intraabdominal pressure parameters were collected from receivers outside..
  Interventions: Other: EXERCISE TRAINING WITHOUT MEDICATION
- Swimming group: The ten participants who are expertise of swim and strong core muscle usage. After ingest the capsule, the signal transmission and intraabdominal pressure parameters were collected from receivers outside..
  Interventions: Other: EXERCISE TRAINING WITHOUT MEDICATION

INTERVENTIONS:
Other: EXERCISE TRAINING WITHOUT MEDICATION — After ingesting the capsular sensor, the participants were request to perform exercise packages and monitor the change of signal transmission rate and shift of intraabdominal pressure level.

SUMMARY:
To test the diagnostic efficacy of using the PressureDOT, an in-body real-time pressure-sensing smart capsule, in monitoring elevated intra-abdominal pressure in subjects.

This study aims to evaluate the PressureDOT (abbreviated as PDT, serial number: PD01), a state-of- the-art continuous pressure sensing system that is among the most advanced in the world. Unlike traditional methods of monitoring intra-abdominal pressure, such as indirectly measuring abdominal pressure by infusing saline into the bladder, PDT offers a minimally invasive, wireless solution intended to reduce the common risk of urinary tract infections associated with traditional methods and significantly decrease the need for manual operations.

The PDT capsule utilizes high-density circuit board technology and is protected by a unibody encapsulation that shields its internal components. This design enables the capsule to precisely and continuously monitor intra-abdominal pressure and temperature while transmitting data to an external receiving device wirelessly. Additionally, the external receiver is equipped with a special algorithm that can instantly track the capsule's speed of movement through the gastrointestinal tract, providing richer data support for clinical diagnosis.

Considering that elevated intra-abdominal pressure is a potential early high-risk factor for various diseases and closely related to the user's health status, this project plans to conduct a Phase I clinical trial across a broad spectrum of groups, including athletes, astronauts, vocalists, individuals undergoing rehabilitation, and any participants at risk of increased intra-abdominal pressure. These groups may face a risk of elevated intra-abdominal pressure due to their unique circumstances. Through this clinical trial, we hope to validate the effectiveness of PDT in the early diagnosis of elevated intra-abdominal pressure, reduce the long-term risk of exposure to high intra-abdominal pressure for participants, and further alleviate the burden on medical practitioners, thereby reducing medical costs.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants without previous surgical history

Exclusion Criteria:

* previous abdominal surgical history
* GI obstruction history
* no need of magnetic resonance imaging in two weeks after capsule ingestion.
* history of swallowing difficulty, dysphagia, odynophagia.

Ages: 20 Months to 65 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The exercise expertises who can ingest capsules without swelling difficulty and can cooperate the monitoring procedure. The age must be above 20 years.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Safety passage of capsule | 7days
  monitor the passage rate of each participants and evaluate the risk for capsule retained rate.

SECONDARY OUTCOMES:
Signal transmission of capsule | 2 days
  The pressure monitoring data transmission rate. We will collect all the signals from participants and calculate the data lost rate.
Intraandominal pressure monitoring | 2 days
  The intraabdominal pressure were record when the capsule stay in the participants' body

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University &Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] de Gennaro JD, de Gennaro CK, Shaw JM, Petelenz TJ, Nygaard IE, Hitchcock RW. The Relationship Between Intra-Abdominal Pressure and Body Acceleration During Exercise. Female Pelvic Med Reconstr Surg. 2019 May/Jun;25(3):231-237. doi: 10.1097/SPV.0000000000000523. PMID 29135811
- [Result] Dietze-Hermosa M, Hitchcock R, Nygaard IE, Shaw JM. Intra-abdominal Pressure and Pelvic Floor Health: Should We Be Thinking About This Relationship Differently? Female Pelvic Med Reconstr Surg. 2020 Jul;26(7):409-414. doi: 10.1097/SPV.0000000000000799. PMID 32574030